CLINICAL TRIAL: NCT06314087
Title: Individualized Tumor Neoantigen Peptide Vaccine in Combination with Unusual Immune Stimulating Radiotherapy in Refractory Solid Tumors (iNATURE) - a Phase II Randomized and Crossover Study
Brief Title: Individualized Neoantigen Therapy with Unusual Radiotherapy Enhancement (iNATURE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Neoantigen Radiotherapy
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Advanced Tumors
Keywords: Neoantigen Peptide Vaccines

STUDY DESIGN:
Masking Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm: Arm #1 (Active Comparator)
  Interventions: Other: Placebo + conventional treatment including radiotherapy
- Experimental arm: Arm #2 (Experimental): Personalized tumor peptide vaccine + conventional treatment including radiotherapy group
  Interventions: Combination Product: Radiation: Radiation Therapy；Biological: Personalized tumor peptide vaccine

INTERVENTIONS:
Other: Placebo + conventional treatment including radiotherapy — Placebo + conventional treatment including radiotherapy
  Other Names: Chemical: per standard care
  Arms: Control arm: Arm #1
Combination Product: Radiation: Radiation Therapy；Biological: Personalized tumor peptide vaccine — The peptide vaccine treatment will take 5 months as a treatment course until the treatment suspension event as stipulated in the plan occurred.
  Arms: Experimental arm: Arm #2

SUMMARY:
In this study, the investigators provide an individualized tumor neoantigen peptide vaccine in combination with radiotherapy to patients with advanced malignant solid tumors. The investigators observe the post-treatment tumor burden status, the immune response induced by immune preparations, and the prolongation of patient survival time, aiming to evaluate the effectiveness and safety of the individualized tumor neoantigen peptide vaccine in combination with radiotherapy

DETAILED DESCRIPTION:
In this study, we intend to recruit patients with advanced tumors that have failed standard treatment or progressed, and conduct a clinical study of individualized tumor neoantigen peptide vaccine combined with radiotherapy according to the process shown in the figure below: (1) for operable patients, tumor tissues were obtained surgically with peripheral blood as the control, and for inoperable patients, tumor tissues were obtained by biopsy with peripheral blood as the control, and DNA was extracted and whole exome sequencing was performed to accurately detect the tumor gene mutation. (2) Confirm the expression of the mutation in the tumor by transcriptome sequencing; (3) Analyze the HLA typing of the patient by exon sequencing results; (4) Integrate the information of mutation, gene expression and HLA typing, predict the binding ability of the mutation with HLA molecules by software, and screen the tumour neoantigen. Tumor neoantigens; in this project, for the same data, three teams will be used to perform neoantigen prediction analysis and validate each other, and the neoantigen sequence with the best solution (intersection of the three teams) will be obtained by combining the three results. (5) Synthesize tumor neoantigen peptide vaccine based on tumor neoantigen, and verify the safety of tumor neoantigen peptide vaccine by in vitro in vivo test; (6) Subjects will first receive precision radiotherapy treatment, and then enter into individualized tumor neoantigen peptide vaccine clinical trial after one week to prove the safety, feasibility and effectiveness of this combined precision therapy.

ELIGIBILITY:
Inclusion Criteria:

1. male or female
2. age>18 years old
3. with advanced or recurrent malignancies diagnosed by pathology and imaging, who have failed systemic standard therapy or disease progression prior to enrollment and have no effective first-line therapy (for effective therapy, refer to the latest version of the treatment guidelines published by the Chinese Society of Clinical Oncology)
4. have at least one imaging measurable lesion
5. with an expected survival of ≥ 3 months
6. with an ECOG (Eastern Cooperative Oncology Group) score of 0-2
7. have access to sufficient tumor DNA (circulating tumor DNA or tissue samples) for analysis, or have genomic/exonic/transcriptional data from tumor and normal tissues and the data meet the analysis requirements, qualified for tumor neoantigen screening, or have prepared neoantigen peptides from a certified company (GMP)
8. women of childbearing age should have negative pregnancy tests within 7 days prior to enrollment, and have no short-term plans to have children and are willing to take protective measures (contraception or other birth control methods) before and during the clinical trial
9. compliant patients who is and able to follow the study protocol and the follow-up procedures

Exclusion Criteria:

1. No neoantigens detected in the sequencing data.
2. with a history of bone marrow or stem cell transplantation
3. enrolled in other therapeutic clinical trials; clinical trials of Chinese medicine
4. with active bacterial or fungal infections
5. with active HIV (human immunodeficiency virus, human immunodeficiency virus), HCV (hepatitis C virus), HBV (hepatitis B virus), or the herpes virus (except for crusting for more than 4 weeks), or with respiratory viral infections (except for those who have been cured for more than 4 weeks)
6. with asthma, autoimmune disease, immunodeficiency
7. under treatment with immunosuppressive drugs
8. with severe coronary or cerebrovascular disease, or other conditions that concerns the investigator for enrollment
9. have clinical, psychological or social factors affecting informed consent or study implementation
10. have a history of drug or peptide allergy, or allergy to other potential immunotherapies
11. no decision making capacity for civil conduct

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — both male and female
Enrollment: 154 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-08-16 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Visits were conducted at the end (or termination) of each course and at 30, 90, and 120 days after the end of the last course for 4 months
  Number of participants with Adverse Events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Cancer Center Hong Kong University Shenzhen Hospital, Principal Investigator — Municipal hospitals
Locations (2):
- China (2):
  - University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - University of Hong Kong-Shenzhen Hospital, Shenzhen, guangzhou

IPD SHARING:
Plan to Share IPD: No
Publications

REFERENCES:
- [Derived] Zhang Y, Hu YF, Ma L, Wu Y, Chao D, Chen X, Xu Z, Su X, Dai W, Huang J, Fu P, Kong FS. A phase II randomized trial of individualized neoantigen peptide vaccine combined with unusual radiotherapy (iNATURE) in advanced solid tumors-GCOG0028. Front Immunol. 2025 Aug 21;16:1538032. doi: 10.3389/fimmu.2025.1538032. eCollection 2025. PMID 40918097